CLINICAL TRIAL: NCT00309023
Title: A Phase I/II, Ascending Multi-Dose Study of BMS-663513, An Agonistic Anti-CD137 Monoclonal Antibody, Administered Every Three Weeks to Patients With Metastatic or Locally Advanced Solid Malignancies
Brief Title: Study of BMS-663513 in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA186-001
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose escalation (Experimental)
  Interventions: Drug: BMS-663513

INTERVENTIONS:
Drug: BMS-663513 — mg/kg, intravenous (IV), 0.3, 1, 3, 6, 10 or 15 mg/kg, once every 3 weeks (q 3 wks), 12 weeks depending on response

SUMMARY:
This is a Phase I/II, ascending, multi-dose study of BMS-663513, an agonistic anti-CD137 monoclonal antibody, administered every three weeks to patients with metastatic or locally advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score of 0-1.
* Measurable disease.
* Absolute neutrophil count (ANC) >= 1,500 cells/mm3
* Platelet count >= 100K cells/mm3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin <= 1.5 x IULN
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase <= 2.5 x institutional upper limit of normal (IULN)
* Patients with advanced solid malignancies must have melanoma, renal or ovarian carcinoma

Exclusion Criteria:

* History of autoimmune diseases.
* Condition requiring the continued use of systemic or topical steroids or the use of immunosuppressive agents.
* Active/symptomatic brain metastasis.
* History of hepatitis B or C.
* Concurrent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assess Safety (Number and distribution and severity adverse events) of subjects | Active treatment of a minimum of 3 months up until disease progression or toxicity; and long-term follow-up to assess time to progression or death will conclude 2 years after the last treatment with BMS-663513.

SECONDARY OUTCOMES:
Efficacy by evaluation of tumor response | At week 12 and every 6 weeks thereafter. Follow-up up to 2 years after last dose of study drug
Assess pharmacokinetic parameters deriving from serum concentration versus time data | Cycle 1 Day 1, Cycle 2 Day 1 and 28, Cycle 3 Day 1 and 8, and Day 1 of every cycle the subject is on study from Cycle 4 and greater; and at study discharge.
Assess pharmacodynamic and immune response analysis | up to 60 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (6):
  - City Of Hope National Medical Center, Duarte, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Local Institution, Toronto, Ontario, Canada
- France (4):
  - Local Institution, Bordeaux
  - Local Institution, Paris
  - Local Institution, Saint-Herblain
  - Local Institution, Villejuif